CLINICAL TRIAL: NCT06776744
Title: EMpower Parents: Effectiveness of EMDR Treatment for Parental PTSD Related to Their Child's Medical Condition: a Randomized Controlled Trial
Brief Title: EMpower Parents: Effectiveness of EMDR Treatment for Parental PTSD Related to Their Child's Medical Condition.
Acronym: EMpower
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Lotte Haverman, Head of Pediatric Psychology Research Section, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL85854.018.24
Record Dates: First submitted 2024-12-23; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: All Acute Pediatric Conditions; All Chronic Pediatric Conditions
Keywords: EMDR; Pediatrics; Posttraumatic stress; Parental PTSD; Parents; Trauma therapy; E-health
MeSH Terms: interventions — Eye Movement Desensitization Reprocessing; Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EMDR in person (Experimental): For both intervention conditions (EMDRip and EMDRr), short EMDR treatment, 4 x 1.5 hour divided over 2 half-days, will be offered following the standard eight-phase protocol (14). Parents in the EMDRip condition will receive EMDR treatment at the Emma Children's Hospital.
  Interventions: Other: Eye Movement Desensitization and Reprocessing (EMDR)
- EMDR remote (Experimental): For both intervention conditions (EMDRip and EMDRr), short EMDR treatment, 4 x 1.5 hour divided over 2 half-days, will be offered following the standard eight-phase protocol (14). Parents in the EMDRr condition will receive EMDR treatment remote via the online web-based tool EMDR platform.
  Interventions: Other: Eye Movement Desensitization and Reprocessing (EMDR)
- Waiting list (No Intervention)

INTERVENTIONS:
Other: Eye Movement Desensitization and Reprocessing (EMDR) — Eye Movement Desensitization and Reprocessing (EMDR) treatment. EMDR is one of the first-choice evidence based treatments for PTSD. During an EMDR session, the traumatic memory is brought to the surface including associated images, thoughts, feelings and body sensations, while simultaneously focusing on an external distracting stimulus (e.g., lateral eye movements).
  Other Names: Psychological intervention
  Arms: EMDR in person; EMDR remote

SUMMARY:
The goal of this clinical trial is to learn if short EMDR treatment offered in two modalities (face to face and remote) is effective in reducing PTSD symptoms and comorbid symptoms for parents of children with diverse chronic and acute medical conditions.

The main question is:

• Is short EMDR treatment effective in reducing PTSD symptoms in parents of children with chronic or acute medical conditions?

Researchers will compare in person and remote EMDR treatment to a waiting list group to see if the treatment is effective.

Participants in the intervention conditions will participate in four in person or remote EMDR sessions, each lasting 1.5 hours, spread across two half-days. Participants in the waiting list condition will receive this treatment after a period of 3 months.

DETAILED DESCRIPTION:
Objective: The primary objective is to assess the effectiveness of a brief (two half-day) in person (EMDRip) and remote (EMDRr) EMDR therapy compared to control group in reducing posttraumatic stress symptoms in parents of children with a chronic or acute medical condition.

The secondary objectives are to assess the effectiveness of brief EMDRip and EMDRr for parents of children with a severe chronic or acute medical condition 1) in reducing psychological comorbidity in parents (psychopathology in general: Depression, Anxiety, and Somatization, and parenting stress), 2) in reducing posttraumatic stress symptoms of their child with a chronic or acute medical condition, and 3) in improving relationship quality between the parent and spouse and between the parent and the child with a severe chronic or acute medical condition. 4) To evaluate the feasibility of EMDRip versus EMDRr.5) To describe the traumatic experiences and future worries (targets) the parents of children with a severe chronic or acute medical condition struggle with.

Study design: This study will be a randomized controlled trial with three study arms: in person EMDR (EMDRip), remote EMDR (EMDRr), waiting list (Control).

Intervention: The EMDR intervention in this study consists of four in person or remote EMDR sessions, each lasting 1.5 hours, spread across two half-days, approximately one week will elapse between the two treatment days. EMDR treatment will be offered by licensed therapists at Amsterdam UMC.

ELIGIBILITY:
Inclusion Criteria:

* One of the three conditions below on the PTSD Check List for DSM-5 (PCL-5): A 'moderately or higher' (2-4) score for at least one symptom in each cluster (B, C, D or E), or Three of the four PTSD criteria (one B symptom, one C symptom, two D symptoms and two E symptoms), or A (sub) clinical total score (>24).
* Being motivated for brief EMDR treatment.
* Parenting a child under treatment of a healthcare provider at the Emma Children's Hospital, Amsterdam UMC.
* Having sufficient knowledge of the Dutch language to complete the questionnaires.

Exclusion Criteria:

* Major interfering acute medical or psychiatric condition, such as psychosis, substance dependence or high risk for suicide.
* Insufficient fluency of the Dutch language.
* Receiving psychological trauma treatment by another therapist at the same time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic stress (symptoms) assessed with the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | From T0 [enrolment] to T1 [2 weeks post end of treatment]

SECONDARY OUTCOMES:
Psychological comorbidity - Anxiety assessed with the Dutch-Flemish PROMIS Bank v1.0 - Anxiety | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Psychological comorbidity - Depression assessed with the Dutch-Flemish PROMIS Item Bank v1.0 - Depression | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Psychological comorbidity - Somatization assessed with the Brief Symptom Inventory-18, BSI-18, subscale Somatic Symptoms | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Parenting stress assessed with the Parenting Burden Questionnaire, OBVL | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Parent-child relationship assessed with the Parenting Burden Questionnaire, OBVL | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Distress assessed with the Distress Thermometer for Parents, DT-P | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Trauma symptoms child assessed with the Child and Adolescent Trauma Screen, CATS, 3-6 and 7-17 parent version, based on the DSM-5 criteria for PTSD | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Social support assessed with the Social Support subscale of the Family Questionnaire, GVL | From T0 [enrolment] to T1 [2 weeks post end of treatment]
Partner relationship assessed with the Partner Relationship subscale of the Family Questionnaire, GVL | From T0 [enrolment] to T1 [2 weeks post end of treatment]

OTHER OUTCOMES:
Feasibility, self-composed questionnaire | 2 weeks post treatment follow-up (T1ip, T1r, T.1.c)
  To assess the feasibility of EMDR in person versus EMDR remote
Therapy preference, self-composed question | Tscreen: part of the first set-of questionnaires parents complete to check for eligibility, pre-intervention.
  To assess potential therapy preference (in person, remote or hybrid) before start of treatment
New traumatic experiences during treatment, self-composed question | At every follow-up measurement moment: T1c: 6 weeks post T0 follow-up, T2c: 16 weeks post T0 follow-up, T1ip, T1r, T1.1c: 2 weeks post end of treatment, T2ip, T2r, T2.1c: 3 months post end of treatment, T3ip, T3r: 6 months post end of treatment.
  To assess if new traumatic experiences occurred after treatment ended
Further treatment need, self-composed question | At the last measurement moment for each group: T3ip, T3r: 6 months post end of treatment T2.1c: 3 months post end of treatment
  To assess if participants are in need for psychological treatment after the EMDR treatment of the study
Intake data: traumatic experiences and future worries | At the psychological intake (in between baseline measurement and the start of the intervention)
  During the psychological intake, the following data is collected: 1) Complaints parents, 2) Information about child's illness, 3) Targets (traumatic experiences): title, short description, child's age, SUD (memory), intrusion, frequency, 4) Mental video check/future template, 5) Other information, 6) Psychoeducation PTSD, 7) Explanation EMDR and practice round, 8) Date, time and location of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Haverman, Dr., Principal Investigator — Amsterdam UMC

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vesseur EM, de Roos C, Scholten L, Haverman L. EMpower Parents: Effectiveness of EMDR treatment for parental PTSD related to a child's medical condition in a randomized controlled trial. BMC Psychol. 2025 Jul 17;13(1):799. doi: 10.1186/s40359-025-03043-x. PMID 40676651